CLINICAL TRIAL: NCT00092157
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Study to Evaluate the Tolerability and Efficacy of the Co-Administration of Simvastatin 20 mg/Day and Fenofibrate 160 mg/Day Compared to Simvastatin 20 mg/Day Alone for 12 Weeks of Treatment in Patients With Combined Hyperlipidemia-Simvastatin and Fenofibrate Efficacy Trial (SAFARI)
Brief Title: Effectiveness of Two Approved Drugs in Lowering High Cholesterol (0733-224)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0733-224; 2004_060
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: High cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0733, simvastatin
Drug: Comparator: simvastatin

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of two approved drugs in lowering high cholesterol when taken together, compared to taking only one of the drugs.

DETAILED DESCRIPTION:
The duration of treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Elevated cholesterol level

Exclusion Criteria:

* Liver disease
* Known allergies to study drugs

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2002-05-01 (Actual); Primary Completion 2003-03-03 (Actual); Study Completion 2003-03-04 (Actual)

PRIMARY OUTCOMES:
Fasting triglyceride levels at 12 weeks.

SECONDARY OUTCOMES:
Total Cholesterol, LDL-C, HDL-C, VLDL-C, VLDL-TG, Apo A-I, and Apo B, CRP, PAI-1, fibrinogen, fasting plasma glucose, and fasting insulin

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Grundy SM, Vega GL, Yuan Z, Battisti WP, Brady WE, Palmisano J. Effectiveness and tolerability of simvastatin plus fenofibrate for combined hyperlipidemia (the SAFARI trial). Am J Cardiol. 2005 Feb 15;95(4):462-8. doi: 10.1016/j.amjcard.2004.10.012. PMID 15695129
- [Background] Grundy SM, Vega GL, Tomassini JE, Tershakovec AM. Correlation of non-high-density lipoprotein cholesterol and low-density lipoprotein cholesterol with apolipoprotein B during simvastatin + fenofibrate therapy in patients with combined hyperlipidemia (a subanalysis of the SAFARI trial). Am J Cardiol. 2009 Aug 15;104(4):548-53. doi: 10.1016/j.amjcard.2009.04.018. PMID 19660610